CLINICAL TRIAL: NCT01800123
Title: Continuous EtCO2 Monitoring in Acute Self Poisoned Patients Admitted in an Emergency Department
Brief Title: EtCO2 Monitoring in Acute Self-poisoning
Acronym: CAPNOTOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-14
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Acute Intentional Overdose
Keywords: Intoxication, overdose, poisoning, EtCO2, emergency medicine
MeSH Terms: conditions — Drug Overdose; Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute poisoning: Consecutive acute drug self poisoned patients admitted in the ED.

SUMMARY:
There is no consensus on monitoring criteria in acute self poisoning. Clinical scores, vital signs or lactatemia have failed to prove good predictive value.

The main acute self poisoning complication is decreased consciousness level with consequent increased risk of hypoxemia and aspiration pneumonitis.

Several clinical studies have recently shown that EtCO2 monitoring can be valuable in procedural sedation in the emergency department. It is able to predict hypoxemia before any SaO2 decrease and any complications related to these procedures.

We therefore hypothesized that EtCO2 could help in acute self poisoning patients' monitoring in the ED.

ELIGIBILITY:
Inclusion Criteria:

* >18y/o
* acute self poisoning patients
* patients requiring monitoring according to physician's opinion
* patients not requiring invasive ventilation at ED admission

Exclusion Criteria:

* Pregnant woman
* patients deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18y/o admitted in the ED for acute self poisoning.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
ROC curve of maximal EtCO2 to predict poisoning complication | During the first 2 hours of ED admission
  Poisoning complications are defined as:
  Hypoxia (Spo2<93%) and/or Respiratory rate <10/min or >25/min and/or ICU admission and/or Oro tracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Genoble university hospital, Grenoble, France

REFERENCES:
- [Derived] Viglino D, Bourez D, Collomb-Muret R, Schwebel C, Tazarourte K, Dumanoir P, Paquier C, Danel V, Debaty G, Maignan M. Noninvasive End Tidal CO2 Is Unhelpful in the Prediction of Complications in Deliberate Drug Poisoning. Ann Emerg Med. 2016 Jul;68(1):62-70.e1. doi: 10.1016/j.annemergmed.2015.11.037. Epub 2016 Jan 23. PMID 26810758